CLINICAL TRIAL: NCT05801731
Title: A Decentralized Study on Dietary Influences on Cognitive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Responsible Party: Principal Investigator, Jeroen Schmitt, Senior Principal Investigator, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2022-059
Record Dates: First submitted 2023-03-09; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Glucose Metabolism; Cognitive Function
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study will be carried out according to a decentralized, randomized, placebo controlled, double-blind, cross-over design.
Who Masked: Participant, Investigator
Masking Description: The randomization list will be prepared by an independent staff who is not part of the current study. A non-speaking code will be used for each of the snack types. The study team members will be kept blinded to the order of snack given to the participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Low-GI snack, administered at 10.00 and 16.00 during the test days
  Interventions: Other: Intervention
- Control (Active Comparator): Normal GI snack, administered at 10.00 and 16.00 during the test days
  Interventions: Other: Control

INTERVENTIONS:
Other: Intervention — The low GI snack is a biscuit with a Glycemic Index of 23.8 ± 3.3. The low GI snack contains plain flour, fibre, plant-based protein, vegetable oil and a low GI sweetener.
  The interventional snacks (control, experimental) are matched for caloric content.
  Arms: Experimental
Other: Control — The normal GI snack is a biscuit with a Glycemic Index of 54.4 ± 6.3. The control snack is formulated using basic ingredients for a biscuit recipe consisting of all-purpose flour, butter, sugar, vanilla flavour, baking soda, egg and salt.
  Arms: Control

SUMMARY:
The current study aims to investigate the cognitive effects of diet-induced blood glucose fluctuations on cognitive performance in healthy older adults over multiple days, taking advantage of the currently available techniques to continuously measure blood glucose levels and to assess cognitive performance in a real-life setting.

In this fully decentralized study, subjects will undergo two times a three-day measurement period, where their blood glucose will be continuously measured by a minimally invasive sensor and where the cognitive performance is measured at multiple time points throughout a day using a short test battery administered on their mobile phone. In addition to receiving standardized breakfast and lunch meals, the subjects are administered a low-GI(Glycemic Index) or normal-GI(Glycemic Index) snack in the morning and afternoon.

DETAILED DESCRIPTION:
The study has two main scientific objectives. First, the investigators aim to investigate the acute effect of a low versus high-GI snack taken mid-morning or mid-afternoon on cognition, appetite, alertness and mood. To this end the investigators will compare the pre-snack and ~2-hour snack measurements of the two snacks. The investigators hypothesize that the low-GI(Glycemic Index) snack, due to a blunted and sustained PPGR, leads to better cognition, appetite and alertness ratings. Secondly, the investigators aim to explore how daily fluctuations in blood glucose are associated with cognition, mood, appetite and alertness in healthy older adults. To this end the investigators will conduct exploratory correlational analyses between blood glucose parameters, the behavioural outcomes, and subject characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 - 65 years
* Own and use a smartphone that is capable to run the study applications (Android 4.4 or later, OS 12.0 or later)
* Adequate fluency in the English language to understand the inform consent process, study instructions and study assessments
* Sufficient vision and hearing to complete study procedures based on medical judgment
* Willing and able to participate and to give written consent to comply with study procedures

Exclusion Criteria:

* Presence or history of a metabolic, neurological, or psychiatric disease
* Use of prescription or OTC medication that may influence gastrointestinal, metabolic or neurological functioning
* Any health, functional or lifestyle factor that in the judgement of the investigator may interfere with the ability to comply with study procedures and/or the generation of valid study data
* Known food allergies
* Use of illicit drugs
* Alcohol intake >1 units/day • BMI <18.5 or >30 kg/m²
* Are a member of the research team or their immediate family members. Immediate family member is defined as spouse, parent, child, or sibling, whether biological or legally adopted

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Spatial working Memory | 6 test days
  Spatial working memory is measured using Dot Memory Task. During the task, participants are presented with a set of dots on a mobile screen for a brief period of time. Following a short delay, a second set of dots is presented, and participants are asked to determine whether any of the dots in the second set were also present in the first set. Participants respond by pressing a button to indicate whether the second set of dots was a match or a non-match to the first set. The task typically involves varying the number of dots in each set to determine the participant's working memory capacity. The primary outcomes are accuracy(%) and reaction speed in milliseconds.

SECONDARY OUTCOMES:
Subjective Cognitive ability | 6 test days
  On a Visual Analog Scale that ranges from 0 to 100, where 0 represents "Not at all" and 100 indicates "Very Much," the answer to the question regarding one's cognitive ability, "'I am feeling mentally sharp," is obtained.
Subjective Alertness | 6 test days
  On a Visual Analog Scale that ranges from 0 to 100, where 0 represents "Not at all" and 100 indicates "Very Much," the answer to the question regarding one's alertness, "I am feeling tired," is obtained.
Subjective Mood | 6 test days
  On a Visual Analog Scale that ranges from 0 to 100, where 0 represents "Not at all" and 100 indicates "Very Much," the answer to the question regarding one's mood, "I am feeling relaxed," is obtained.
Subjective Appetite | 6 test days
  On a Visual Analog Scale that ranges from 0 to 100, where 0 represents "Not at all" and 100 indicates "Very Much," the answer to the question regarding one's appetite, "I am feeling hungry," is obtained.
Blood Glucose | 11 days
  Blood glucose is measured continuously through Freestyle Libre CGM (Continuous Glucose Monitor) for 11 days
Speed of processing | 6 test days
  The speed of processing is measured using the Symbol Search Task. The task involves presenting participants with pairs of symbols on a screen and requiring them to match these pairs with other pairs displayed at the top of the screen. Two pairs of symbols are presented at the bottom of the screen, and participants are asked to quickly determine which of the two pairs matches the pairs displayed at the top of the screen. The task measures the median reaction time (in milliseconds) of correctly matched symbol pairs. Participants are given a brief interval of 200 milliseconds between each response and the following stimulus to complete the task. This task is used to assess how quickly individuals can process visual information and make accurate decisions.
Sustained attention | 6 Test days
  Sustained attention is measured using a 3-min Psychomotor Vigilance Task (PVT). The outcome variables are the median reaction time (ms) of valid responses and the number of lapses (reaction time exceeding 500ms).

OTHER OUTCOMES:
HBA1c | Day 0, Prior the actual test
  HbA1c test is a simple blood test that measures your average blood sugar levels over the past 3 months. It's one of the most commonly used tests to diagnose prediabetes and diabetes. HbA1c is measured in two units of measurement: mmol/mol and percent (percentage of total hemoglobin)

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Schmitt, PhD, Principal Investigator — Senior Principal Investigator
Locations (1):
- Singapore Institute for Clinical Trials, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez-Bueno C, Martinez-Vizcaino V, Lopez EJ, Visier-Alfonso ME, Redondo-Tebar A, Cavero-Redondo I. Comparative Effect of Low-Glycemic Index versus High-Glycemic Index Breakfasts on Cognitive Function: A Systematic Review and Meta-Analysis. Nutrients. 2019 Jul 24;11(8):1706. doi: 10.3390/nu11081706. PMID 31344892
- [Background] Philippou E, Constantinou M. The influence of glycemic index on cognitive functioning: a systematic review of the evidence. Adv Nutr. 2014 Mar 1;5(2):119-30. doi: 10.3945/an.113.004960. PMID 24618754
- [Derived] Mohapatra L, Cabral R, Bhatnagar M, Chan PW, Ng M, Chua XY, Soon CS, Massar S, de Iorio M, Schmitt JAJ. Glucoregulatory status modulates acute cognitive effects of repeated low-glycaemic snack consumption in older adults: a decentralized randomized controlled trial. Eur J Nutr. 2025 May 26;64(5):189. doi: 10.1007/s00394-025-03712-y. PMID 40419805

DOCUMENTS (1):
  • Informed Consent Form (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/31/NCT05801731/ICF_000.pdf